CLINICAL TRIAL: NCT00359853
Title: Randomized Double-Blid Placebo Controlled Trial Assessing Norfloxacin In The Primary Prophylaxis Of Spontaneous Bacterial Peritonitis In Advanced Cirrhosis
Brief Title: Norfloxacin In The Primary Prophylaxis Of Spontaneous Bacterial Peritonitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 00-pbe-mnjf-2
Record Dates: First submitted 2006-08-01; First posted 2006-08-03 (Estimated); Last update posted 2006-08-03 (Estimated); Status verified 2004-06

CONDITIONS: Spontaneous Bacterial Peritonitis; Hepatorenal Syndrome; Cirrhosis
Keywords: Norfloxacin, primary prophylaxis, SBP
MeSH Terms: conditions — Hepatorenal Syndrome; Fibrosis | interventions — Norfloxacin

INTERVENTIONS:
Drug: Oral norfloxacin

SUMMARY:
Advanced liver disease and low ascitic fluid protein concentration have been identified as risk factors for spontaneous bacterial peritonitis in cirrhosis. Moreover, renal impairment and hyponatremia increase mortality rate of this infection. Aims: To investigate if oral administration of norfloxacin prevents the first episode of SBP, hepatorenal syndrome and improves survival in cirrhotic patients with ascites and low protein concentration in ascitic fluid (<15 g/L) and at least one of the following inclusion criteria: functional renal failure (serum creatinine ≥ 1,2 mg/dl or BUN ≥ 25 mg/dl), hyponatremia (serum sodium ≤ 130 mEq/L) or advanced liver disease (Child ≥ 9 points with serum bilirubin ≥ 3 mg/dl). Methods: Prospective, multicenter, randomized, double-blind placebo controlled trial comparing oral norfloxacin (400 mg/d; n=35) with placebo (n=35).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years, protein concentration in ascitic fluid < 15 g/L and at least one of the following: serum creatinine ≥ 1.2 mg/dl or BUN ≥ 25 mg/dl, serum sodium ≤ 130 mEq/L or severe liver failure as defined by a Child-Pugh score ≥ 9 points and a serum bilirubin ≥ 3 mg/dl.

Exclusion Criteria:

* Previous history of spontaneous bacterial peritonitis or of norfloxacin prophylaxis, allergy to quinolones, hepatocellular carcinoma, organic renal failure and HIV infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2000-09; Study Completion 2005-03

PRIMARY OUTCOMES:
Short-term and long-term survival

SECONDARY OUTCOMES:
Prevention of the first episode of spontaneous bacterial peritonitis
Prevention of hepatorenal syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Miquel Navasa, MD, Principal Investigator — Liver Unit. Hospital Clinic Barcelona
Locations (1):
- Hospital Clinic Barcelona, Barcelona, Catalonia, Spain